CLINICAL TRIAL: NCT02130661
Title: A Phase I, Two-part, Open-label Study to Evaluate the Pharmacokinetics of Rilapladib (SB-659032) and Its Metabolites, and to Determine the Effect of Repeat Dose Itraconazole on the Pharmacokinetics of Rilapladib in Healthy Volunteers
Brief Title: Study to Determine the Effect of Itraconazole on the Pharmacokinetics of Rilapladib (SB659032) in Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201274
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Alzheimer's Disease
Keywords: drug interaction; healthy volunteer; rilapladib; SB-659032; Alzheimer's disease; itraconazole
MeSH Terms: conditions — Alzheimer Disease | interventions — rilapladib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Subjects will receive 250 mg of rilapladib once daily (QD) for 14 days (Days 1-14)
  Interventions: Drug: Rilapladib 250 mg
- Part B (Experimental): Subjects will receive 25 mg of rilapladib QD for 1 day (Day 1), 200 mg of itraconazole twice daily (BID) for 1 day (Day 8) and QD for 2 days (Days 9-10). Subjects will receive 25 mg of rilapladib + 200 mg of itraconazole for 1 day (Day 11) and 200 mg of itraconazole QD for 6 days (Day 12-17)
  Interventions: Drug: Rilapladib 25 mg; Drug: Itraconazole

INTERVENTIONS:
Drug: Rilapladib 25 mg — White, round, biconvex, film coated tablet of 25 mg. Taken orally along with food.
  Arms: Part B
Drug: Rilapladib 250 mg — White, round, biconvex, film coated tablet of 250 mg. Taken orally along with food.
  Arms: Part A
Drug: Itraconazole — 100 mg capsule with a blue opaque cap and pink transparent body. Taken orally along with food.
  Arms: Part B

SUMMARY:
Rilapladib is a potent and selective inhibitor of lipoprotein associated phospholipase A2 (Lp-PLA2), which was previously under development for the treatment of atherosclerosis and is currently being developed for the treatment of Alzheimer's disease.

This study is a single-center, open-label, two-part study. The two study parts will run independently. Subjects dosed in one part of this study will not be permitted to participate in the other part.

Part A will investigate the pharmacokinetic profile of rilapladib and its metabolites, SB-664601 and GSK1174379, after single dose and steady state dosing of rilapladib 250 milligram (mg) along with the biliary and urinary elimination pathways of rilapladib 250 mg. Part B will determine the effect of repeat administration of itraconazole on the PK of a single oral dose of rilapladib 25 mg.

Healthy male and female subjects, aged 18-65 years, will be recruited for this study. Ten subjects will be recruited for Part A and 20 subjects will be recruited for Part B.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and Electrocardiogram (ECG). A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the Glaxosmithkline (GSK) Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A subject with an alanine aminotransferase (ALT), alkaline phosphatase or bilirubin laboratory result outside the reference range may be included only if the Investigator and GSK Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-International units/milliliter (MIU/mL) and estradiol < 40 picogram (pg)/mL (<147 picomole/Litre [pmol/L]) is confirmatory].
* Body weight >= 50 kilogram (kg) and body mass index (BMI) within the range 19-32 kg/square meter (m^2) (inclusive).
* Based on single QT duration corrected for heart rate by Fridericia's formula (QTcF): QTcF <450millisecond (msec); or QTcF <480 msec in subjects with right bundle branch block.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

Criteria Based Upon Medical History

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), or prior cholecystectomy.
* History of asthma, anaphylaxis or anaphylactoid reactions, or severe allergic responses.
* Lifetime history of suicide attempt or active suicidal ideation within the past six months.
* Current major depressive episode or a previous episode of depression requiring medical intervention.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinical research unit uses heparin to maintain intravenous cannula patency).
* History of sensitivity to compounds with a chemical structure related to rilapladib or itraconazole, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Any contraindications for itraconazole administration.
* Requiring the use of oral or injectable strong Cytochrome P450 3A4 (CYP3A4) inhibitors or use of other CYP3A4 inhibitors/inducers within 14 days prior to dosing.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.

Criteria Based Upon Diagnostic Assessments

* A positive pre-study Hepatitis B surface antigen, positive Hepatitis C antibody result, or positive test for Human Immunodeficiency Virus (HIV) antibody.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug or alcohol screen.

Other Criteria

* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Previous participation in this study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices within 7 days prior to the first dose of study medication until collection of the final pharmacokinetic sample.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax), time of occurrence of Cmax (Tmax), area under the concentration-time curve over the dosing interval (AUC(0-Tau)) of rilapladib parent compound after single and repeat dosing, in part A of the study. | Day (D)1: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24 hours (hrs) post-dose, and D14: pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 32, 48 (D16), 96 (D18), 144 (D20), 240 (D24) and 336 (D28) hrs post-dose. Pre-dose on Days 11, 12 and 13
  Cmax, Tmax and AUC (0-Tau) will be used to evaluate the pharmacokinetics of rilapladib after single and repeat dosing of rilapladib 250 mg.
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity)), and terminal phase half-life (T1/2) of rilapladib after repeat dosing, in part A of the study | D1: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24 hrs post-dose, and D14: pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 32, 48 (D16), 96 (D18), 144 (D20), 240 (D24) and 336 (D28) hrs post-dose. Pre-dose on Days 11, 12 and 13
  AUC(0-infinity) and T1/2 of rilapladib will be used to evaluate the pharmacokinetics of rilapladib and its metabolites after repeat dosing of rilapladib 250 mg.
Cmax, Tmax, AUC(0-tau), and area under the concentration-time curve from time zero (pre-dose) to time of last quantifiable concentration (AUC(0-t)) of SB-664601 and GSK1174379 after single and repeat dosing, in part A of the study | D1: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24 hrs post-dose, and D14: pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 32, 48 (D16), 96 (D18), 144 (D20), 240 (D24) and 336 (D28) hrs post-dose. Pre-dose on Days 11, 12 and 13
  Cmax, Tmax, AUC(0-tau), and AUC(0-t) will be used to evaluate the pharmacokinetics of SB-664601 and GSK1174379 after single and repeat dosing of rilapladib 250 mg.
AUC(0-infinity) and T1/2 of SB-664601 and GSK1174379 after repeat dosing, as data permit, in part A of the study. | D1: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24 hrs post-dose, and D14: pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 32, 48 (D16), 96 (D18), 144 (D20), 240 (D24) and 336 (D28) hrs post-dose. Pre-dose on Days 11, 12 and 13
  AUC(0-infinity) and T1/2 will be used to evaluate the pharmacokinetics of SB-664601 and GSK1174379 after repeat dosing of rilapladib 250 mg.
AUC(0 infinity), AUC(0 t), and Cmax of rilapladib alone and in the presence of itraconazole in part B of the study. | D1 : Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 32, 48 (D3), 96 (D5), 144 (D7) hours post dose, and on D 11: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 32, 48 (D13), 96 (D15), 144 (D17) hours post dose
  AUC(0 infinity), AUC(0 t), and Cmax will be used to evaluate the effect of repeat oral dosing of itraconazole on the pharmacokinetics of single dose rilapladib 25 mg.

SECONDARY OUTCOMES:
Safety and tolerability of repeat oral doses of rilapladib 250 mg assessed by adverse events (AEs), in part A of the study. | Up to Day 38
  AEs will be collected from the start of Study Treatment and until the follow-up
Safety and tolerability of repeat oral doses of rilapladib 250 mg assessed by 12-lead electrocardiogram (ECG) parameters, in part A of the study. | Up to Day 38
  Single 12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures pulse rate (PR), QRS, QT, and QTcF intervals.
Safety and tolerability of repeat oral doses of rilapladib 250 mg assessed by measuring vital signs, in part A of the study. | Up to Day 38
  Vital sign measurements will be performed in semi-supine or supine position after 10 minutes rest and will include systolic and diastolic blood pressure and pulse rate.
Safety and tolerability of repeat oral doses of rilapladib 250 mg assessed by laboratory tests, in part A of the study. | Up to Day 38
  Laboratory tests will include haematology, clinical chemistry, urinalysis and additional parameters.
Tmax and T1/2 of rilapladib alone and in the presence of itraconazole, in part B of the study. | D1 : Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 32, 48 (D3), 96 (D5), 144 (D7) hours post dose, and on D 11: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 32, 48 (D13), 96 (D15), 144 (D17) hours post dose
  Tmax and T1/2 will be used to evaluate the effect of repeat oral dosing of itraconazole on the secondary PK parameters of rilapladib 25 mg.
AUC(0-infinity), AUC(0-t), Cmax, Tmax and T1/2 of rilapladib metabolites, SB-664601 and GSK1174379, alone and in the presence of itraconazole, in part B of the study. | D1 : Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 32, 48 (D3), 96 (D5), 144 (D7) hours post dose, and on D 11: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 32, 48 (D13), 96 (D15), 144 (D17) hours post dose
  AUC(0-infinity), AUC(0-t), Cmax, Tmax and T1/2 will be used to evaluate the effect of repeat oral dosing of itraconazole on the PK of the rilapladib metabolites, SB-554601 and GSK1174379, after single dose of rilapladib 25 mg.
Safety and tolerability of single oral dose of rilapladib 25 mg when dosed alone and concomitantly with itraconazole, assessed by AEs, in part B of the study. | Up to Day 27
  AEs will be collected from the start of Study Treatment and until the follow-up
Safety and tolerability of single oral dose of rilapladib 25 mg when dosed alone and concomitantly with itraconazole, assessed using ECG parameters, in part B of the study. | Up to Day 27
  Single 12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals.
Safety and tolerability of single oral dose of rilapladib 25 mg when dosed alone and concomitantly with itraconazole, assessed as vital signs, in part B of the study. | Up to Day 27
  Vital sign measurements will be performed in semi-supine or supine position after 10 minutes rest and will include systolic and diastolic blood pressure and pulse rate.
Safety and tolerability of single oral dose of rilapladib 25 mg when dosed alone and concomitantly with itraconazole, assessed by laboratory tests, in part B of the study. | Up to Day 27
  Laboratory tests will include haematology, clinical chemistry, urinalysis and additional parameters.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline